CLINICAL TRIAL: NCT02816203
Title: Vacuum Device for Hemostasis in Obstetrics and Gynecology. Feasibility Study for Postpartum Hemorrhage
Brief Title: Vacuum Device for Hemostasis in Obstetrics and Gynecology
Acronym: HEMOGYN2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); HEMOSQUID (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC15.060
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Primary Postpartum Hemorrhage; Administration of Sulprostone; Vaginal Childbirth
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary Hemostatic Intra-Uterine suction cup (Experimental): Patients who present primary postpartum hemorrhage requiring administration of Nalador and the suction cup placed in the uterine cavity
  Interventions: Device: Hemostatic Intra-Uterine suction cup

INTERVENTIONS:
Device: Hemostatic Intra-Uterine suction cup — The hemostatic intra-uterine suction cup is introduced to the uterine cavity and a negative pressure is applied into the device.

SUMMARY:
Postpartum hemorrhage (PPH), is the leading cause of maternal mortality and is responsible for approximately 25% of maternal mortality deaths.It is defined as blood loss in excess of 500 ml following vaginal childbirth. Primary (immediate) PPH occurs within the first 24 hours after delivery.

In clinical practice, if after giving birth, the placenta is not expelled naturally, an active management should be triggered. After obstetric maneuvers therapeutic, options begin with uterotonic treatments before considering invasive treatments such as embolization, vessel ligation and hysterectomy. However, the morbidity associated with these techniques and the desire to preserve fertility mean that new therapeutic solutions have been conceived, which has recently led to the development of an innovative intrauterine hemostasis medical device : a hemostatic intrauterine suction cup.

Assuming that postpartum hemorrhages are mainly due to uterine atony, we propose in this biomedical research, the study of a new medical device. Our hypothesis is that the uterine walls will append to the walls of the suction cup after the latter is put under vacuum. The actuation of the suction cup will lead to the aspiration of all sides of the uterus.

Considering that postpartum haemorrhage is an emergency situation where vital prognosis of the patient is engaged, we selected to collect the consent of the patient using an emergengy procedure.

DETAILED DESCRIPTION:
In this study, as a first pass in human of this innovative non CE marked medical device, we aim to demonstrate the feasibility of using the hemostatic intrauterine suction cup for patients who present primary PPH (blood loss ≥ 500ml) after a vaginal delivery requiring administration of Nalador®. We will evaluate the placement of hemostatic suction cup in the uterus, the application of vacuum and its removal from the uterus.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 45 years old
* patient under loco-regional anesthesia
* patient who presents primary postpartum hemorrhage (blood loss ≥ 500ml) after a vaginal childbirth requiring administration of Nalador®.
* affiliation to the French social security system or equivalent
* patient who has signed a consent to participate

Exclusion Criteria:

* patient with a uterine malformation
* patient allergic to silicon
* patient under general anesthesia
* patient who delivered via caesarean section
* patient with fever or suspected infection during labor
* person deprived of freedom by judicial or administrative decision
* person hospitalized without their consent
* person under legal protection
* person hospitalized for psychiatric care

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the feasibility of using the hemostatic intrauterine suction cup in patients who present primary PPH (blood loss ≥ 500ml) after a vaginal childbirth requiring the administration of Nalador®. | 36 month
  The primary outcome is composite and consists of 3 the following component outcomes:
  1. Qualification of success or failure of the introduction of the suction cup in the uterine cavity
  2. Qualification of success or failure to create negative pressure in the suction cup. The negative pressure is validated if vacuum is maintained for at least 30 seconds.
  3. Qualification of success or failure of removing the suction cup in its entirety.
  The feasibility of using the suction cup will be validated if success is obtained for the 3 component outcomes.

SECONDARY OUTCOMES:
Evaluation of the ease of the placement of the suction cup by the clinician | 36 month
  Visual quantitative satisfaction scale
Evaluation of whether the bleeding stops after each time the suction cup is put under vacuum. For each patient, the cup may be put once or twice under vacuum. | 36 month
  Subjective evaluation of whether bleeding stops by the clinician after each time the suction cup is put under vacuum.
Evaluation of the ease of removal of the suction cup by the clinician | 36 month
  Visual quantitative satisfaction scale
Quantification of blood loss during delivery | 36 month
  Volume of blood collected in the container of the pump and in the collection bag from the beginning of the delivery until the removal of the suction cup
Evaluation of the number of patients for whom invasive treatment is necessary in order to stop the bleeding | 36 month
  Number of patients for whom embolization or surgery is indicated
Assessment of the duration of time required to place and remove the suction cup | 36 month
  Time duration for the placement and removal of the suction cup

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Equy, MD, Principal Investigator — Clinic of Gynecology and Obstetrics, University Hospital Grenoble, France
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No